CLINICAL TRIAL: NCT06372769
Title: Comparative Analysis of Myoelectric Activity and Mandibular Movement in Healthy and Temporomandibular Disorder Subjects
Brief Title: Myoelectric Activity and Mandibular Movement for the Diagnosis of Temporomandibular Disorder
Status: Completed | Type: Observational
Sponsor: Stomatological Hospital Affiliated with Fujian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 20240304
Record Dates: First submitted 2024-04-12; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Temporomandibular Disorder
Keywords: Temporomandibular joint disorder;; Surface electromyography;; Mandibular kinematics;; Sex difference;; Diagnosis.
MeSH Terms: conditions — Temporomandibular Joint Disorders; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy young adults with individual normal occlusion: Healthy subjects who fulfilled the following criteria: centred midline and no marked restriction and deviation of mouth opening and closing; overjet and overbite of 1-3 mm, bilateral molar support with molar and cusp relation of Angle's class I, and presence of complete permanent dentition, except third molars.
  Interventions: Diagnostic Test: electromyograph and kinesiograph
- Temporomandibular disorder patients with disc displacement: Patients with unilateral or bilateral temporomandibular joint (TMJ) disc displacement symptoms, such as TMJ clicking, TMJ locking, and limitation in opening mouth were included in the study. The study did not cover the patients with muscle disorders (myofascial pain), with arthralgia, osteoarthritis, and osteoarthrosis, with TMJ fracture, with dentofacial deformity, with systemic disease affecting TMJ, and undergone TMD treatments.
  Interventions: Diagnostic Test: electromyograph and kinesiograph

INTERVENTIONS:
Diagnostic Test: electromyograph and kinesiograph — The sEMG of the anterior temporalis (TA), masseter (MM), sternocleidomastoid (cervical group, CG), and digastric (DA) were recorded simultaneously with an sEMG device (K7/EMG, USA) using disposable silver/silver chloride bipolar surface electrodes.
  First, sEMG was conducted on four pairs of muscles (TA, MM, CG, and DA) in the MPP, and subjects were guided to maintain the face and jaw as relaxed as possible. To determine the relative efficiency of muscle function, the second test was performed to measure the sEMG of TA and MM during the maximal biting force against natural dentition. In the third test, subjects were guided to clench three times to monitor early motor unit recruitment as they closed from rest through freeway space to initial tooth contact.
  Kinesiographic recordings were performed using a kinesiograph (K7/Computerized Mandibular Scanning (CMS), USA) that measured the maximum mouth opening (MMO) and opening and closing velocities.

SUMMARY:
This study aimed to provide normal reference values of surface electromyography (sEMG) and mandibular kinematics in Chinese young adults, compare the sex differences and assess the diagnosis value of these indices.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) are one of the leading causes of craniofacial pain, and a high incidence of TMD in young adults has been reported. Previous studies have used sEMG and mandibular kinematic analysis to diagnose TMD. This was an observational study that healthy young adults with individual normal occlusion were strictly selected by diagnosis standard, and TMD patients with disc displacement were recruited. The sEMG signals of the anterior temporalis (TA), masseter (MM), and sternocleidomastoid and digastric were recorded in the mandibular postural positions (MPP) and during maximal voluntary clenching (MVC) with K7 electromyograph. Mandibular kinematics, including maximum opening and opening/closing velocities, were assessed by K7 kinesiograph.

ELIGIBILITY:
Inclusion Criteria:

* Centred midline and no marked restriction and deviation of mouth opening and closing; ·Overjet and overbite of 1-3 mm, bilateral molar support with molar and cusp relation of Angle's class I;
* Presence of complete permanent dentition, except third molars.

Exclusion Criteria:

* History of local or general trauma;
* Presence of systemic diseases, neurological or psychiatric disorders, muscular diseases, cervical pain, or TMD based on the Research Diagnostic Criteria (RDC);
* Pregnancy;
* Consumption of anti-inflammatory, analgesic, antidepressant, or myorelaxant drugs;
* Presence of parafunctional facets and anamnesis of parafunctional tooth clenching, bruxism, or unilateral chewing;
* Presence of obvious dentition crowding or spacing, malposed, supernumerary or fractured tooth, visible caries, tooth abrasion/hypersensitivity, toothache, periodontal disease, or occlusal discomfort;
* Fixed or removable restorations, tooth filling, or occlusal adjustment that affected the occlusal surfaces;
* Previous or concurrent orthodontic, orthognathic, or TMJ treatment.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers were recruited from college students of Fujian Medical University, while the temporomandibular disorder participants were recruited through public invitations, via recruitment posters and personal contacts.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Surface electromyography (μV) | 3 days
  The sEMG of the anterior temporalis (TA), masseter (MM), sternocleidomastoid (cervical group, CG), and digastric (DA) during mandibular postural position and maximal clench were recorded.

SECONDARY OUTCOMES:
Mandibular kinematics (mm, mm/s) | 3 days
  Kinesiographic recordings were performed using a kinesiograph, the maximum mouth Maximal opening, maximal and average opening and closing velocities were measured.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Stomatological Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xiaojie X, Yiling C, Honglei L, Jiamei P, Xiaoyong W, Hao Y, Hui C. Comparative analysis of myoelectric activity and mandibular movement in healthy and nonpainful articular temporomandibular disorder subjects. Clin Oral Investig. 2024 Oct 21;28(11):605. doi: 10.1007/s00784-024-05957-z. PMID 39428401